CLINICAL TRIAL: NCT04790539
Title: an Single Arm, Single Center Phase II Clinical Study of Shr-1210 Combined With Paclitaxel-albumin and Carboplatin in the First-line Treatment of Extensive Stage Small Cell Lung Cancer
Brief Title: a Study of SHR1210 in Combination With Paclitaxel-albumin and Carboplatin in Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Prof. Caicun Zhou, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-1st-IIT-SHR1210-naP-CB
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — camrelizumab; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+Paclitaxel-albumin+Carboplatin (Experimental): SHR-1210 was given in the first day of each cycle, Carboplatin was given in the first day of each cycle, Paclitaxel-albumin was given in the first day of each cycle, with intravenous drip.
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD-1 IgG4 monoclonal antibody
  Other Names: Anti-PD-1 Antibody

SUMMARY:
This project is to to explore the safety and efficacy of shr-1210 combined with albumin, paclitaxel and carboplatin in the first-line treatment of extensive small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Confirmed diagnosis of Extensive small cell lung cancer
* Eastern Cooperative Oncology Group performance status (PS) of 0 to 1
* The function of vital organs meets the following requirements. WBC ≥ 3.0 × 10^9/L, ANC≥1.5×10^9/L, PLT≥100×10^9/L, Hb≥9g/dL, ALT and AST ≤2.5 times ULN, TBIL ≤1.5 x ULN, CREA ≤1.5 x ULN or CCr≥50mL/min. INR≤1.5 x ULN, APTT ≤1.5 x ULN
* have not received first-line systemic therapy or immunosuppressive therapy for es-sclc
* The estimated survival period is more than 8 weeks
* The subjects voluntarily joined the study, signed informed consent,

Exclusion Criteria:

* Active or untreated CNS metastases were detected by computed tomography (CT) or magnetic resonance imaging (MRI);
* Leptomeningeal diseases
* Uncontrolled or symptomatic hypercalcemia
* Active, known or suspected autoimmune diseases
* have received any T cell co stimulation or immune checkpoint therapy
* Corticosteroids (> 10 mg / day prednisone or equivalent) or other immunosuppressants were used within 14 days before the first dose of study drug
* Subjects had active infections
* Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation
* Known to be allergic to the study drug or excipients, known to have a serious allergic reaction to any kind of monoclonal antibody; have a history of hypersensitivity to Paclitaxel-albumin or Carboplatin
* According to the researcher's judgment, there are other factors that may lead to the termination of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | up to 24 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months
  Determined using RECIST v1.1 criteria
Progression-Free Survival(PFS) | Up to approximately 24 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.
Overall Survival(OS) | Up to approximately 24 months
  Defined as the time from randomization to death from any cause
Number of Subjects with treatment-related adverse events (AEs) | Up to approximately 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI-CTC AE 5.0

IPD SHARING:
Plan to Share IPD: Undecided